CLINICAL TRIAL: NCT05013463
Title: Open-label, Single-center, Single-arm Futility Trial Evaluating the Combination of Oral Hydroxychloroquine 200mg BID and Indapamide 2.5mg OD for Reducing Progression of Disability in People With Secondary Progressive Multiple Sclerosis (SPMS)
Brief Title: Hydroxychloroquine and Indapamide in SPMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCQ_IND_MS01
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Hydroxychloroquine; Indapamide

STUDY DESIGN:
Intervention Model Description: Simon-2-stage MinMax design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxychloroquine and Indapamide (Experimental): Oral Hydroxychloroquine, 200mg BID Oral Indapamide, 2.5 mg OD
  Interventions: Drug: Hydroxychloroquine Pill; Drug: Indapamide Pill

INTERVENTIONS:
Drug: Hydroxychloroquine Pill — Oral Hydroxychloroquine, 200mg BID
  Other Names: Plaquenil
Drug: Indapamide Pill — Oral Indapamide, 2.5 mg OD
  Other Names: Lozol

SUMMARY:
The purpose of this clinical trial is to determine if HCQ in a dose of 400mg daily and indapamide in a dose of 2.5mg daily can help in reducing the progression of disability in people with secondary progressive multiple sclerosis.

The number of participants in this study will be 35. A maximum of 42 people with SPMS will be included. The trial is funded through internal funding through the University of Calgary. There is no sponsorship from any pharmaceutical industry.

DETAILED DESCRIPTION:
In patients with SPMS, there is ongoing slow and continuous loss of nerve cells, which causes damage to the brain and spinal cord. This ultimately becomes noticeable as slowly and continuously worsening disability. While the cause of this ongoing damage is unknown, it appears that at least part of the damage may be caused by cells in the brain called "microglia" (a type of immune cell that resides in the brain and spinal cord). These microglial cells can have beneficial roles, for instance when they clear away debris, but they can also cause damage to brain cells. In SPMS, microglial cells are often found to be in a state of activation, and it is currently believed that this constant activation of microglial cells is likely an important cause of the ongoing damage to brain cells. Another harmful process affecting patients with SPMS is "oxidative stress". Oxidative stress occurs when immune cells in the brain and spinal cord are activated and produce substances that may damage nerve cells. Current treatments for MS mostly are meant to prevent relapses and are beneficial in relapsing-remitting MS, but so far there are no treatments that benefit people with SPMS who do not experience relapses. Better therapies are needed for SPMS, and it is believed that treatments that reduce the activation of microglial cells and oxidative stress may be useful.

The medication Hydroxychloroquine (HCQ) reduces the activity of human microglia in laboratory experiments. Animal experiments also showed that treatment with HCQ reduces disease severity in an animal model of MS. HCQ, therefore, may also reduce the activity of microglia in people with SPMS, and hopefully prevent or slow down the progression of disability in SPMS. HCQ is currently approved in Canada to treat malaria and rheumatic diseases Systemic Lupus Erythematosus (SLE) and Rheumatoid Arthritis (RA). HCQ is available as a tablet that is usually taken two times per day. Doses up to 600mg per are used in clinical practice, but it is estimated that a dose of only 400mg daily, given as two doses of 200mg, will be sufficient to decrease the activity of microglia in patients with SPMS. HCQ is usually well tolerated.

Indapamide (IND) is a medication to treat high blood pressure that can reduce oxidative stress and improve the survival of nerve cells in laboratory studies. IND is currently approved to treat high blood pressure. IND is available in tablet form and is usually taken once a day, the most typical dose is 2.5mg. It is estimated that a dose of 2.5mg per day will be sufficient to treat oxidative stress in SPMS. IND is usually well tolerated.

Following a MinMax Simon-2-stage design, the study will require 35 patients with a complete 18 month follow-up. Presuming 20% drop-out, the investigators anticipate recruiting up to 42 patients. The trial will be conducted as follows: patients will continuously enter into the study until 35 patients have completed 18 months of follow-up with at least 75% adherence which will be measured by study drug count.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Men and women aged 18 and 60 years inclusive
* With SPMS, according to current diagnostic criteria
* Screening Expanded Disability Status Scale score between 4.0 and 6.5 inclusive.
* Screening timed 25-foot walk (average of two trials) of 9 seconds or more

Exclusion Criteria:

* Individuals with retinopathy
* Individuals whose screening ophthalmological exam shows retinopathy
* Individuals with renal insufficiency (pre-existing or developing during the trial)
* Individuals with significant hepatic impairment (pre-existing or developing during the trial)
* Individuals with abnormal screening labs
* Individuals with cardiac arrhythmia
* Individuals with a prolonged QT interval: individuals with frequency corrected QT (QTc) intervals of more than 450ms (men) or 470ms (women) at the screening examination will not be included in the study, and participants with QTc intervals of greater than 500ms on any of the other ECG examinations throughout the study will be excluded from the study.
* Individuals with porphyria
* Individuals with an allergy or other intolerability to HCQ or IND
* Individuals who use Fampridine or 4-aminopyridine
* Individuals who start Fampridine or 4-aminopyridine during the trial
* Individuals who start Baclofen or Tizanidine during the trial
* Individuals who increase the dose of Baclofen or Tizanidine during the trial
* Individuals who receive treatment with Botulinum toxin in the leg muscles during the trial
* Individuals who use siponimod, amiodarone, dapsone, digoxin or antimalarial drugs other than HCQ
* Pregnant or breast-feeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Timed 25-Foot Walk (T25FW) | Change in Timed 25-Foot Walk performance between the 6 month and 18 month visit
  quantitative ambulation performance test

SECONDARY OUTCOMES:
9-Hole Peg Test | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  Brief, standardized, quantitative test of upper extremity
Symbol Digit Modalities Test | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  measures cognitive processing speed and working memory
Functional Systems and Expanded Disability Status Scale (EDSS) | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  Standard measure of neurologic impairment that is used to describe disability in MS. The neurological assessment comprises seven functional system on a scale of 0 (no disability) to 5 or 6 (more severe disability). EDSS steps 5.0 to 9.5 are defined by the impairment to walking.
Modified Fatigue Impact Scale (MFIS) | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  Structured, self-report questionnaire with 21 items concerning how fatigue impact patients quality of life, using a scale that ranges from 0 ("no problem") to 4 ("extreme problem"). Scores are then tallied to produce an overall score with a potential maximum of 160.
Multiple Sclerosis Quality of Life Scale 54 item version | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  54-item multidimensional health-related quality of life measure that combines both generic and MS-specific items

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes